CLINICAL TRIAL: NCT03944408
Title: The Efficacy and Safety of a Metal Bare Stent With 125I Seeds for the Treatment of Malignant Central Airway Compared to a Metal Bare Stent: A Multicentric Randomized Controlled Study.
Brief Title: A Metal Bare Stent With 125 Iodine （125I）Seeds for the Treatment of Malignant Central Airway Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Shanghai 10th People's Hospital (Other); The Second Affiliated Hospital of Xiamen Medical College (Unknown); Anhui Chest Hospital (Other); China Meitan General Hospital (Other); The Second Hospital of Hebei Medical University (Other); West China Hospital (Other); The Second Affiliated Hospital of Fujian Medical University (Other); Wuhan Central Hospital (Other); Wuhan No.1 Hospital (Other); Hunan People's Hospital (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); Yichang Central People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wzchencs
Record Dates: First submitted 2019-05-05; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Malignant Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A metal bare stent with 125I seeds (Experimental): 125I seeds fixed on the metal bare stent, then stent implantation
  Interventions: Procedure: stent implantation
- A metal bare stent (Other): A metal bare stent implantation
  Interventions: Procedure: stent implantation

INTERVENTIONS:
Procedure: stent implantation — stent implantation

SUMMARY:
Malignant central airway stenosis caused by primary or metastatic malignant tumor may lead to dyspnea even death of patients.With the rapid development of interventional pulmonology, bronchoscopic therapy has become the main treatment for malignant central airway stenosis. Metal stent implantation in airway can quickly relieve respiratory obstruction and improve quality of life.However, the tumor tissue can continue to grow into metal stent and obstruct airway again. This is the shortcoming of metal bare stents, which often need further treatment to keep airway open, including ablation, laser, cryotherapy, external radiotherapy or systemic anti-tumor drug therapy.Metal stent implantation combined with external radiotherapy can effectively reduce the incidence of airway restenosis.However, complications of external radiotherapy are high, including bone marrow suppression, radioactive pneumonia, radioactive esophagitis, myocardial injury and tracheoesophageal fistula, of which may cause serious consequences and even cause death of the patient.125I radioactive seeds have been one of the mature radioactive interventional therapy, which release X rays, and γ rays. Because of the short radioactive distance, 125I seeds can destruct tumor cells in tumor site and promote apoptosis and necrosis of tumor cells around the obstruction of the airway, meanwhile cause little damage to the surrounding normal tissues. Some studies showed that 125I seed implantation of lung tumor lesions achieved good short-term results.Therefore, the investigators hypothesize that 125I seeds fixed on the metal bare stent can not only improve the patient's breathing difficulties, but also play a role in killing tumor cells. At present, there have been reports of related clinical cases and monocentric control studies of malignant central airway stenosis treated with the implantation of metal stent with 125I seeds, but there is a lack of multicentric clinical studies with large samples.

DETAILED DESCRIPTION:
It is an open, multicentric randomized controlled clinical trial conducted in China, and plan to recruiting 200 patients who suffer malignant central airway stenosis. To evaluate the efficacy and safety of metal stent with 125I seeds group and metal bare stent group in the treatment of malignant central airway stenosis, follow-up should be done within 1 week, 1 month, and 3 months after the first treatment, followed by every 3 months. The contents include review of bronchoscopy and chest CT, blood routine, immune indicators (IgA, immunoglobulin M（Ig M）, IgG), evaluation of general conditions. The patients of the first group need emission-computed tomography（ECT） imaging or positron emission tomography-computed tomography （PET-CT） examination within 1 month. If the patient has severe dyspnea, emergency bronchoscopy should be performed .

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-75 years old, male or female who is not pregnant
2. Comply with the diagnosis of malignant central airway stenosis, and undergo chest CT or bronchoscopy to confirm that the stenosis degree is above 50% and need to be implanted with airway metal stent; or the patient has obvious dyspnea due to airway stenosis, obstructive pneumonia
3. Subjects voluntarily joined the study and signed informed consent, with good compliance and follow-up.
4. Unable or refused surgery
5. Unable or refused external radiation therapy
6. Unable or refuse systemic tumor-related drugs therapy within 3 months

Exclusion Criteria:

1. The distal end of the stenosis is unpredictable, and the stent treatment may not be satisfactory;
2. Severe arrhythmia, acute myocardial ischemia, uncontrollable hypertensive crisis;
3. Severe coagulopathy
4. Severe organ dysfunction (except respiratory insufficiency)
5. Allergic to anesthetics
6. Airway fistula lesions
7. The narrow lesion involves 2cm inside the glottis
8. History of extrathoracic radiation therapy in the past 6 months
9. Severe myelosuppression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
stenosis grade | the first month after stent implantation
  Stenosis grade was classified as 5 grades on the cross-sectional CT imaging area: grade 0
  = non-appreciable stenosis; grade 1, 2, 3, and 4 = 25, 50, 75, and 90% decrease in area, respectively; grade 5 = complete obstruction
stenosis grade | the third month after stent implantation
  Stenosis grade was classified as 5 grades on the cross-sectional CT imaging area: grade 0
  = non-appreciable stenosis; grade 1, 2, 3, and 4 = 25, 50, 75, and 90% decrease in area, respectively; grade 5 = complete obstruction

SECONDARY OUTCOMES:
overall survival （OS） | From randomization until death （up to 24 months）
  overall survival
technical success | one week after stent implantation
  successful implantation of the stent across the stricture with appropriate positioning of the stent and full expansion
complications and side effects | From randomization until death （up to 24 months）
  Possible radiation related complications included neutropenia, decrease in IgA, IgG, and IgM, and leakage of radioactive seeds.Neutropenia was defined as a total white blood cell count b4000/mm3 in the plasma. The leakage of radioactive seeds was defined as the detection of non-target radioactive source verified by radiography
tumor growth rate | From randomization until death （up to 24 months）
  the size of tumor assessed by CT after stent implantation
the time of emergency endoscopic treatment | From randomization until death （up to 24 months）
  record the time of emergency endoscopic treatment for the recurrent severe dyspnea of patient

CONTACTS AND LOCATIONS:
Overall Officials: Chengshui Chen, doctor, Study Chair — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The first affiliated hospital of wenzhou medical university, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ernst A, Feller-Kopman D, Becker HD, Mehta AC. Central airway obstruction. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1278-97. doi: 10.1164/rccm.200210-1181SO. PMID 15187010
- [Result] Ong P, Grosu HB, Debiane L, Casal RF, Eapen GA, Jimenez CA, Noor L, Ost DE. Long-term quality-adjusted survival following therapeutic bronchoscopy for malignant central airway obstruction. Thorax. 2019 Feb;74(2):141-156. doi: 10.1136/thoraxjnl-2018-211521. Epub 2018 Sep 25. PMID 30254139
- [Result] Wood DE, Liu YH, Vallieres E, Karmy-Jones R, Mulligan MS. Airway stenting for malignant and benign tracheobronchial stenosis. Ann Thorac Surg. 2003 Jul;76(1):167-72; discussion 173-4. doi: 10.1016/s0003-4975(03)00033-x. PMID 12842534
- [Result] Saad CP, Murthy S, Krizmanich G, Mehta AC. Self-expandable metallic airway stents and flexible bronchoscopy: long-term outcomes analysis. Chest. 2003 Nov;124(5):1993-9. doi: 10.1378/chest.124.5.1993. PMID 14605078
- [Result] Sabath BF, Ost DE. Update on airway stents. Curr Opin Pulm Med. 2018 Jul;24(4):343-349. doi: 10.1097/MCP.0000000000000486. PMID 29538079
- [Result] Lemaire A, Burfeind WR, Toloza E, Balderson S, Petersen RP, Harpole DH Jr, D'Amico TA. Outcomes of tracheobronchial stents in patients with malignant airway disease. Ann Thorac Surg. 2005 Aug;80(2):434-7; discussion 437-8. doi: 10.1016/j.athoracsur.2005.02.071. PMID 16039180
- [Result] Rochet N, Hauswald H, Schmaus M, Hensley F, Huber P, Eberhardt R, Herth FJ, Debus J, Neuhof D. Safety and efficacy of thoracic external beam radiotherapy after airway stenting in malignant airway obstruction. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):e129-35. doi: 10.1016/j.ijrobp.2011.11.055. PMID 22516383
- [Result] Qu A, Wang H, Li J, Wang J, Liu J, Hou Y, Huang L, Zhao Y. Biological effects of (125)i seeds radiation on A549 lung cancer cells: G2/M arrest and enhanced cell death. Cancer Invest. 2014 Jul;32(6):209-17. doi: 10.3109/07357907.2014.905585. Epub 2014 Apr 18. PMID 24745612
- [Result] Wang Y, Lu J, Guo JH, Zhu GY, Zhu HD, Chen L, Wang C, Teng GJ. A Novel Tracheobronchial Stent Loaded with 125I Seeds in Patients with Malignant Airway Obstruction Compared to a Conventional Stent: A Prospective Randomized Controlled Study. EBioMedicine. 2018 Jul;33:269-275. doi: 10.1016/j.ebiom.2018.06.006. Epub 2018 Jun 14. PMID 29909977
- [Result] Lu M, Pu D, Zhang W, Liao J, Zhang T, Yang G, Liu Z, Singh S, Gao F, Zhang F. Trans-bronchoscopy with implantation of 125I radioactive seeds in patients with pulmonary atelectasis induced by lung cancer. Oncol Lett. 2015 Jul;10(1):216-222. doi: 10.3892/ol.2015.3204. Epub 2015 May 13. PMID 26171002
- [Result] Mallick I, Sharma SC, Behera D. Endobronchial brachytherapy for symptom palliation in non-small cell lung cancer--analysis of symptom response, endoscopic improvement and quality of life. Lung Cancer. 2007 Mar;55(3):313-8. doi: 10.1016/j.lungcan.2006.10.018. Epub 2006 Dec 8. PMID 17157949
- [Result] Wang Y, Guo JH, Zhu GY, Zhu HD, Chen L, Lu J, Wang C, Teng GJ. A Novel Self-Expandable, Radioactive Airway Stent Loaded with 125I Seeds: A Feasibility and Safety Study in Healthy Beagle Dog. Cardiovasc Intervent Radiol. 2017 Jul;40(7):1086-1093. doi: 10.1007/s00270-017-1639-8. Epub 2017 Apr 7. PMID 28389860